CLINICAL TRIAL: NCT06321094
Title: Vericiguat in Patients With Acute Coronary Syndrome and Reduced Ejection Fraction: The EVE-ACSrEF Study
Brief Title: Effect of Vericiguat on Acute Coronary Syndrome( ACS）Patients With Ejection Fraction <45%
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: EVE-ACSrEF
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndrome; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who take vericiguat: Grouped by their treatment preference, some of ACS patients with ejection fraction(EF)<45% are to take vericiguat.
- patients who donot take vericiguat: Grouped by their treatment preference, some of ACS patients with ejection fraction(EF)<45% arenot to take vericiguat.

SUMMARY:
Investigators evaluate whether differences exsit in acute coronary syndrome（ACS） patients with ejection <45% between participants who take vericiguat regularly and those who donot.

DETAILED DESCRIPTION:
Vericiguat, a novel soluble guanylate cyclase stimulator, reduced the incidence of cardiovascular death or hospitalization for HF in a population of high-risk patients with heart failure with reduced ejection fraction （HFrEF ）who had recently been hospitalized or received intravenous diuretic therapy.Given the increasing incidence of patients with ACS and its challenges posing to life，investigators intend to conduct a prospective observational study. Investigators choose several meaningful endpoints including the time of cardiovascular death or heart failure（HF) hospitalization、inflammatory markers、the value of N-terminal pro-B-type natriuretic peptide(NT-proBNP)、results of echocardiogram and life quality score.By collecting these datas and work on a group of analysis ，investigators evaluate whether differences exsit in ACS patients with ejection <45% between participants who take vericiguat regularly and those who donot.

ELIGIBILITY:
Inclusion Criteria:

* 1.Provide written informed consent for the trial.
* 2.Has acute coronary syndrome (unstable angina, non-ST elevation myocardial infarction [NSTEMI], or ST elevation myocardial infarction [STEMI]) or coronary revascularization (coronary artery bypass grafting [CABG] or percutaneous coronary intervention [PCI]).
* 3.ejection fraction <45%.
* 4.Be male or female, aged greater than18 and less than 90 on the day of signing informed consent.

Exclusion Criteria.

* 1.SBP<100mmHg.
* 2.Is pregnant or breastfeeding or plans to become pregnant or to breastfeed during the course of the trial.
* 3.Has severe hepatic insufficiency or renal insufficiency.
* 4.Has malignancy or other non-cardiac condition limiting life expectancy to <1 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
a composite of death from cardiovascular causes or first hospitalization for heart failure | from baseline to one year

SECONDARY OUTCOMES:
results of echocardiogram | from baseline to one year
  changes in left ventricular ejection fraction during the follow-up
the numerical value of NT-proBNP | from baseline to one year
  an important biomarker of heart failure
life quality score | from baseline to one year
  Investigators choose Kansas City Cardiomyopathy Questionnaire(KCCQ) to evaluate life quality of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong PW, Pieske B, Anstrom KJ, Ezekowitz J, Hernandez AF, Butler J, Lam CSP, Ponikowski P, Voors AA, Jia G, McNulty SE, Patel MJ, Roessig L, Koglin J, O'Connor CM; VICTORIA Study Group. Vericiguat in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2020 May 14;382(20):1883-1893. doi: 10.1056/NEJMoa1915928. Epub 2020 Mar 28. PMID 32222134
- [Result] Saldarriaga C, Atar D, Stebbins A, Lewis BS, Abidin IZ, Blaustein RO, Butler J, Ezekowitz JA, Hernandez AF, Lam CSP, O'Connor CM, Pieske B, Ponikowski P, Roessig L, Voors AA, Anstrom KJ, Armstrong PW; VICTORIA Study Group. Vericiguat in patients with coronary artery disease and heart failure with reduced ejection fraction. Eur J Heart Fail. 2022 May;24(5):782-790. doi: 10.1002/ejhf.2468. Epub 2022 Mar 20. PMID 35239245
- [Result] Ponikowski P, Alemayehu W, Oto A, Bahit MC, Noori E, Patel MJ, Butler J, Ezekowitz JA, Hernandez AF, Lam CSP, O'Connor CM, Pieske B, Roessig L, Voors AA, Westerhout C, Armstrong PW; VICTORIA Study Group. Vericiguat in patients with atrial fibrillation and heart failure with reduced ejection fraction: insights from the VICTORIA trial. Eur J Heart Fail. 2021 Aug;23(8):1300-1312. doi: 10.1002/ejhf.2285. Epub 2021 Jul 18. PMID 34191395
- [Result] Chen T, Kong B, Shuai W, Gong Y, Zhang J, Huang H. Vericiguat alleviates ventricular remodeling and arrhythmias in mouse models of myocardial infarction via CaMKII signaling. Life Sci. 2023 Dec 1;334:122184. doi: 10.1016/j.lfs.2023.122184. Epub 2023 Oct 20. PMID 37866806